CLINICAL TRIAL: NCT06329596
Title: Periodontal Disease and Alterations in the Oral and Vaginal Microbiome Communities Among Gravidae Chewing Xylitol-gum in Malawi: Microbiome Alterations With Xylitol (MAX) in Pregnancy Trial.
Brief Title: Microbiome Alterations With Xylitol (MAX) in Pregnancy
Acronym: MAX
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); University of Washington (Other); Baylor College of Medicine Children's Foundation Malawi (Unknown)
Responsible Party: Principal Investigator, Benjamin Chimarioff Shayo, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-55146; D43TW012274 (NIH)
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Dysbiosis; Inflammation Gum; Placenta-mediated Pregnancy Complications; Microbioata; Neurodevelopmental Changes (Childhood, Ageing)
Keywords: microbial alterations; xylitol; Malawi; infant neurodevelopment
MeSH Terms: conditions — Dysbiosis; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, data collectors (i.e. dental officers, study staff members, clinical officers), and data analysts will be blinded (triple-blinded) to group allocation throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Xylitol gum (Experimental): Participants will receive 6.36grams of daily xylitol; Epic dental gum, 1.06 grams Xylitol per piece of gum; to chew two pieces for 5 minutes after meals, thrice a day.
  Interventions: Dietary Supplement: Xylitol gum
- Sorbitol gum (Placebo Comparator): Participants will receive Epic sorbitol-containing gum (0 grams xylitol/day); to chew two pieces for 5 minutes after meals, thrice a day.
  Interventions: Dietary Supplement: Sorbitol gum

INTERVENTIONS:
Dietary Supplement: Xylitol gum — Two pieces of xylitol gum after meals, thrice a day.
  Other Names: Epic Xylitol gum
  Arms: Xylitol gum
Dietary Supplement: Sorbitol gum — Two pieces of sorbitol gum after meals, thrice a day.
  Arms: Sorbitol gum

SUMMARY:
The purpose of this study is to understand if chewing xylitol-gum initiated before 20 weeks of pregnancy and continued until delivery affects the bacteria that are found in the oral and vaginal cavities, signs of inflammation within the gingiva of the oral cavity, the health of the tissues in the mouth (clinical parameters of periodontal disease) and placentae, and the bacteria in the mouth and gut of newborns among pregnant individuals in Malawi. In addition, we will evaluate the impact of xylitol-containing chewing gum use during pregnancy on the offsprings neurodevelopment at approximately 6- and 18-months corrected age.

DETAILED DESCRIPTION:
After consenting to the study, pregnant participants who have a singleton gestation and are <20 weeks' gestation will be randomised into either the intervention arm ( 6.36grams of daily xylitol; Epic dental gum, 1.06 grams Xylitol per piece of gum; chew two pieces for 5 minutes after meals, thrice a day) or the placebo control arm (Sorbitol Gum base; Epic sorbitol-containing gum, 0 grams/day of xylitol; chew two pieces for 5 minutes after meals, thrice a day) by randomly picking from a group of opaque, sealed envelopes containing group allocation. The participants will also undergo a dental assessment and sampling, and vaginal sampling at enrolment, 28- 30 weeks of pregnancy, at birth - 48 hours and 4-6 weeks after birth. In addition, placental and breastmilk specimens will be obtained at the time of delivery, and stored in a biobank for future analyses. The investigators will also obtain oral and meconium (and stool at 4-6 weeks) samples of their newborns at birth and 4-6 weeks after birth. Furthermore, at 6- and 18-months corrected age, the infants will undergo neurodevelopmental assessments using the the Hammersmith Infant Neurologic Exam (HINE), Developmental Assessment of Young Children 2nd Edition (DAY-C), and Malawi Development Assessment Tool (MDAT). The assessments will be done by two community health workers trained in these methods and will be compared to assessments by a paediatric neurologist.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent. For those under 18 years of age, consent will additionally be sought from the parent or guardian.
* A singleton at <20 weeks' gestation (based on ultrasound or best obstetric measurement)
* Planning to deliver at Area 25 health center.
* Willing to chew two pieces of gum thrice daily for 5 minutes after the morning, day and evening meals throughout pregnancy.
* Willing to undergo at least two dental exams including oral microbiota sampling at study enrolment <20 weeks of pregnancy, 28-30 weeks, at delivery/within 48 hours and 4-6 weeks after giving birth.
* Willing to have at least two vaginal sampling at study enrolment <20 weeks of pregnancy, 28-30 weeks, at delivery/within 48 hours and 4-6 weeks after giving birth.
* Able to speak Chichewa or English.
* Cognitively aware enough to be able to participate in the study.
* Willing to consent to all required aspects of protocol including allowing collection of placenta specimens, infant oral swab and meconium/stool sampling at birth/within 48 hours and 4-6 weeks after.

Exclusion Criteria:

* Those who upon screening and enrolment but dislike the taste of the gum and state they will not chew the gum throughout pregnancy.
* Gravidae with known or suspected non-viable pregnancy (including life threatening congenital anomalies such as cardiac, neurological or others).
* Pregnant individual has a life-threatening diagnosis such as cancer requiring treatment during pregnancy.
* Pregnant women with a known or suspected morbidly adherent placenta (such as placenta accrete, increta and percreta).

Ages: 12 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Periodontal disease at 28-30 weeks of pregnancy | Enrolment and 28-30 weeks of pregnancy.
  The investigators will create scaled periodontal disease score comprising of sum of scores for gingival bleeding (+1 if bleeding was present, per tooth), gingival pockets (+1 for pockets of 4-5 mm and +2 for 6 mm or deeper, per tooth), and loss of attachment (+1 for 4-5 mm loss, +2 for 6-8 mm, +3 for 9-11 mm, and +4 for 12 mm or more, per tooth with values recorded for index teeth) divided by the number of teeth present will be created for every dental visit. A score of >0 will indicate presence of periodontal disease. The investigators will compare periodontal disease status at 28-30 weeks of pregnancy to that at enrolment.

SECONDARY OUTCOMES:
Periodontal disease at 6 weeks postpartum | Enrolment and 6 weeks postpartum
  The investigators will create scaled periodontal disease score comprising of sum of scores for gingival bleeding (+1 if bleeding was present, per tooth), gingival pockets (+1 for pockets of 4-5 mm and +2 for 6 mm or deeper, per tooth), and loss of attachment (+1 for 4-5 mm loss, +2 for 6-8 mm, +3 for 9-11 mm, and +4 for 12 mm or more, per tooth with values recorded for index teeth) divided by the number of teeth present will be created for every dental visit. A score of >0 will indicate presence of periodontal disease. The investigators will compare periodontal disease status at 6 weeks postpartum to that at enrolment.
Alterations in the maternal oral microbiome communities | Enrolment and at 28-30 weeks, delivery and 4-6 weeks after
  Using 16S rRNA sequencing to assess strain level changes in sub gingival plaque composition within and between those exposed to xylitol and placebo gum using exact amplicon sequence variants.
Alterations in the maternal vaginal microbiome communities | Enrolment and at 28-30 weeks, delivery and 4-6 weeks after
  Using 16S rRNA sequencing to assess strain level changes in the vaginal microbiome at the vaginal introitus and posterior fornix. The investigators will compare compositional differences between sites in relationship to treatment
Inflammatory mediator changes in the maternal gingival crevicular fluid compared to changes in the placenta. | Enrolment and at 28-30 weeks, and at delivery
  The investigators will assess changes in local oral inflammation associated with xylitol exposure or not by evaluating the gingival crevicular fluid using a 10-plex pro inflammatory cytokine panel.
Alterations within the infants' oral microbiome communities | 4-6 weeks
  The investigators will us 16S rRNA sequencing to assess strain level changes within the oral swabs of the infants born during the MAX trial and assess changes in the composition within and between those exposed to xylitol and placebo gum.
Alterations within the infants' gut microbiome communities | 4-6 weeks
  The investigators will use 16S rRNA sequencing to assess strain level changes in the stool/meconium samples from the infants' gut microbiome and assess compositional changes within and between those exposed to xylitol and placebo gum.
To determine the impact of chewing xylitol-containing gum (6.4 grams/day) vs placebo gum in pregnancy on neurodevelopmental outcomes of offspring at 6 and 18 months | At 6- and 18- months of corrected age.
  We will use the MDAT z-score as a primary outcome. Secondary outcomes include DAYC-2 raw score and HINE optimality scores and asymmetries. Relevant descriptive statistics, and non-parametric tests will be used in analysis.
To determine whether the addition of the DAYC-2 and HINE to the MDAT at 6 months of age improves the predictive validity for any NDD (1 SD below normative score on any MDAT domain), identified on the MDAT, DAYC-2 and/or HINE at 18 months corrected age. | 6- and 18-months of corrected age
  We will utilise logistic regression to establish a predictive model for addition of the DAYC-2 and HINE to MDAT for NDD at 18 months corrected age.
(Exploratory) To assess the intra-class correlation between an intensively trained Community Health Workers (CHW) in administering the MDAT, DAYC-2, and HINE as compared to a gold-standard examiner (Malawi-based Pediatric Neurologist). | 6- and 18-months corrected age.
  We will use standard measures including Cronbach's alpha coefficient to compare all assessments between CHW and the gold standard examiner and generate a Bland-Altman plot. We will use the results of this exploratory aim to inform a power calculation for a planned future large investigation to determine how many assessments are needed by two examiners to assess the reliability of CHW exams.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Shayo, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Area 25 Health Center, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared for investigators who have an IRB approved project and approach the researchers with a research plan that is approved by the study team.
Supporting Information: Study Protocol
Time Frame: 1 year after the study conclusion will the data become available and be available for approximately 10 years after study completion.
Access Criteria: Investigators interested in the study data should contact the Study PI (Dr. Ben Shayo - Benjamin.shayo@bcm.edu) or study team members (i.e. Dr. Greg Valentine - gcvalent@uw.edu).

REFERENCES:
- [Background] Chen P, Hong F, Yu X. Prevalence of periodontal disease in pregnancy: A systematic review and meta-analysis. J Dent. 2022 Oct;125:104253. doi: 10.1016/j.jdent.2022.104253. Epub 2022 Aug 20. PMID 35998741
- [Background] Robinson JL, Johnson PM, Kister K, Yin MT, Chen J, Wadhwa S. Estrogen signaling impacts temporomandibular joint and periodontal disease pathology. Odontology. 2020 Apr;108(2):153-165. doi: 10.1007/s10266-019-00439-1. Epub 2019 Jul 3. PMID 31270648
- [Background] Alnasser BH, Alkhaldi NK, Alghamdi WK, Alghamdi FT. The Potential Association Between Periodontal Diseases and Adverse Pregnancy Outcomes in Pregnant Women: A Systematic Review of Randomized Clinical Trials. Cureus. 2023 Jan 1;15(1):e33216. doi: 10.7759/cureus.33216. eCollection 2023 Jan. PMID 36733569
- [Background] Bobetsis YA, Graziani F, Gursoy M, Madianos PN. Periodontal disease and adverse pregnancy outcomes. Periodontol 2000. 2020 Jun;83(1):154-174. doi: 10.1111/prd.12294. PMID 32385871
- [Background] Zhang Y, Feng W, Li J, Cui L, Chen ZJ. Periodontal Disease and Adverse Neonatal Outcomes: A Systematic Review and Meta-Analysis. Front Pediatr. 2022 May 4;10:799740. doi: 10.3389/fped.2022.799740. eCollection 2022. PMID 35601423
- [Background] Iheozor-Ejiofor Z, Middleton P, Esposito M, Glenny AM. Treating periodontal disease for preventing adverse birth outcomes in pregnant women. Cochrane Database Syst Rev. 2017 Jun 12;6(6):CD005297. doi: 10.1002/14651858.CD005297.pub3. PMID 28605006
- [Background] Soderling E, Pienihakkinen K. Effects of xylitol and erythritol consumption on mutans streptococci and the oral microbiota: a systematic review. Acta Odontol Scand. 2020 Nov;78(8):599-608. doi: 10.1080/00016357.2020.1788721. Epub 2020 Jul 7. PMID 32633595
- [Background] Marghalani AA, Guinto E, Phan M, Dhar V, Tinanoff N. Effectiveness of Xylitol in Reducing Dental Caries in Children. Pediatr Dent. 2017 Mar 15;39(2):103-110. PMID 28390459
- [Background] Gudnadottir U, Debelius JW, Du J, Hugerth LW, Danielsson H, Schuppe-Koistinen I, Fransson E, Brusselaers N. The vaginal microbiome and the risk of preterm birth: a systematic review and network meta-analysis. Sci Rep. 2022 May 13;12(1):7926. doi: 10.1038/s41598-022-12007-9. PMID 35562576
- [Background] Loimaranta V, Mazurel D, Deng D, Soderling E. Xylitol and erythritol inhibit real-time biofilm formation of Streptococcus mutans. BMC Microbiol. 2020 Jun 29;20(1):184. doi: 10.1186/s12866-020-01867-8. PMID 32600259
- [Background] Soderling E, Pienihakkinen K, Gursoy UK. Effects of sugar-free polyol chewing gums on gingival inflammation: a systematic review. Clin Oral Investig. 2022 Dec;26(12):6881-6891. doi: 10.1007/s00784-022-04729-x. Epub 2022 Oct 14. PMID 36239787
- [Background] Soderling E, Pienihakkinen K. Effects of xylitol chewing gum and candies on the accumulation of dental plaque: a systematic review. Clin Oral Investig. 2022 Jan;26(1):119-129. doi: 10.1007/s00784-021-04225-8. Epub 2021 Oct 22. PMID 34677696